CLINICAL TRIAL: NCT06887894
Title: EVALUATION OF NEW BIOMARKERS IN THE IDENTIFICATION OF UNSTABLE CAROTID PLAQUE
Brief Title: Biomarkers and Unstable Carotid Plaque
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, TINELLI GIOVANNI, Associate Professor of Vascular Surgery, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 0032543/19
Record Dates: First submitted 2023-03-12; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Carotid Artery Diseases
MeSH Terms: conditions — Carotid Artery Diseases | interventions — Endarterectomy, Carotid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Carotid endarterectomy — Carotid endarterectomy, plaque histological analysis and miRNA expression

SUMMARY:
This prospective study investigated associations between circulating miRNAs and symptomatic and asymptomatic ICAS, carotid plaque morphology and future cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Presence of significant internal carotid artery stenosis referred to carotid artery endarterectomy.
* Age>18 years

Exclusion Criteria:

* Presence of significant internal carotid artery stenosis referred to carotid artery stenting

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with significant internal carotid artery stenosis referred to the Unit of Vascular Surgery of Fondazione Policlinico Gemelli IRCCS Rome for carotid artery endoarterectomy.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
miRNA levels | 30 days
  miRNA levels and plaque vulnerability

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma, RM, Italy

IPD SHARING:
Plan to Share IPD: No